CLINICAL TRIAL: NCT05249530
Title: Comparison of EEG Changes Over Time Following Application of Chiropractic Adjustive Force vs Non-force Simulation
Brief Title: Chiropractic Force Versus Touch
Acronym: FVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: I-0015
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to whether they are receiving an adjustment with force or a non-force stimulation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Force (Experimental): Chiropractic spinal adjustment with force
  Interventions: Other: Chiropractic spinal adjustment
- Touch (Active Comparator): non-force stimulation
  Interventions: Other: Non-force simulation

INTERVENTIONS:
Other: Chiropractic spinal adjustment — Chiropractic spinal adjustment
  Arms: Force
Other: Non-force simulation — Non-force simulation
  Arms: Touch

SUMMARY:
The Life University Center for Chiropractic Research is conducting a research study to better understand the physiologic and brain-based differences between the touch and force components of the chiropractic adjustment. Eligible individuals will either receive a chiropractic adjustment with force or a non-force stimulation. Individuals in the force stimulation group will receive an active spinal adjustment with a handheld instrument called an Activator. Individuals in the non-force stimulation group will have one Activator placed on the spine and another Activator clicked away from the spine. This study is not randomized. The first participant will receive an active spinal adjustment, and the second participant will receive a non-force stimulation at the same locations as the first participant. This pattern repeats until all individuals have been recruited (n=30). Outcome assessments include resting state electroencephalography (EEG), electrocardiography (ECG), and blood pressure. Outcome assessments will be captured prior to the adjustment or non-force stimulation, after the adjustment or non-force stimulation, and one week later. Individuals will also undergo a standard health history and chiropractic physical exam at the start of participation.

ELIGIBILITY:
Inclusion Criteria:

* You are between the age of 18 and 50.
* You have not had a chiropractic adjustment in the past 2 weeks.
* You are not currently receiving care such as acupuncture or physical therapy.
* You are currently not taking any medication that may change your brain patterns.

Exclusion Criteria:

* You do not have a history of recent spinal surgery or trauma.
* You do not have any other health conditions that may prevent you from receive chiropractic care. This could include diagnosed osteoporosis.
* You are not pregnant.
* You do not have a severe mental health condition.
* You do not have a known heart condition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) Power spectrum | Baseline, beginning of the study
  64 channels of EEG will be recorded. A fast Fourier transform will be computed to provide a power spectrum of frequencies 1-50.
Electroencephalography (EEG) Power spectrum | through study completion, an average of 1 year
  64 channels of EEG will be recorded. A fast Fourier transform will be computed to provide a power spectrum of frequencies 1-50.
Electroencephalography (EEG) Power spectrum | One week follow up
  64 channels of EEG will be recorded. A fast Fourier transform will be computed to provide a power spectrum of frequencies 1-50.
Electrocardiogram (ECG) R-R intervals | Baseline, beginning of the study
  Three leads will be placed on the torso to capture a Lead II ECG. R-R intervals will be calculated.
Electrocardiogram (ECG) R-R intervals | through study completion, an average of 1 year
  Three leads will be placed on the torso to capture a Lead II ECG. R-R intervals will be calculated.
Electrocardiogram (ECG) R-R intervals | one-week follow up
  Three leads will be placed on the torso to capture a Lead II ECG. R-R intervals will be calculated.
Blood pressure | Baseline, beginning of the study
  Blood pressure will be captured using an automatic blood pressure cuff
Blood pressure | through study completion, an average of 1 year
  Blood pressure will be captured using an automatic blood pressure cuff
Blood pressure | one-week follow up
  Blood pressure will be captured using an automatic blood pressure cuff

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, PhD, DC, Principal Investigator — Life Univeristy
Locations (1):
- Life University Center for Chiropractic Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No